CLINICAL TRIAL: NCT02677142
Title: A Randomized Control Trial to Evaluate the Efficacy of a Group Social Skills Intervention for Childhood Survivors of Brain Tumours
Brief Title: Evaluating the Efficacy of a Group Social Skills Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Maru Barrera, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000014297
Record Dates: First submitted 2015-12-14; First posted 2016-02-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Brain Tumours
Keywords: pediatric; Childhood Brain Tumour Survivors; Social Skills Rating System; social skills intervention program (SSIP)
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Control Group (CG) (Active Comparator): Behavioural: CG: Social Skills Activities: Participants in this arm will experience an 8-week manualized intervention program with activities and games. Sessions will NOT be designed around a specific social skill and activities and games will NOT have a specific focus. Sessions will be conducted by facilitators who will receive the standard training for volunteers and will work under the supervision of one of the investigators at each site.
  Interventions: Behavioral: CG - social skills activities
- Experimental Group (EG) (Experimental): Behavioral: Structured social skills training program, SSIP. Participants in this arm will experience an 8-week manualized intervention program that addresses six major social skills, one per session, starting with easier skills (Social Initiation and Friendship Making, Cooperation) and moving towards more complex skills (Managing Teasing and Bullying, Conflict Resolution, Empathy, and Assertion). Sessions will be conducted by facilitators who will receive the standard training for volunteers and will work under the supervision of one of the investigators at each site.
  Interventions: Behavioral: Structured social skills training program, SSIP

INTERVENTIONS:
Behavioral: Structured social skills training program, SSIP — Detailed, session by session, in the manual written for this purpose. It addresses six major social skills, one per session, starting with easier skills (Social Initiation and Friendship Making, Cooperation) and moving towards more complex skills (Managing Teasing and Bullying, Conflict Resolution, Empathy, and Assertion).
  Arms: Experimental Group (EG)
Behavioral: CG - social skills activities — Sessions will not be designed around a specific social skill and activities and games will not have a specific focus. CG sessions will be conducted by facilitators who will receive the standard training for volunteers and will work under the supervision of one of the investigators at each site.
  Arms: Attention Control Group (CG)

SUMMARY:
Tumours affecting the brain are a very heterogeneous group of diseases. Accordingly, treatment strategies vary widely depending on child's age, tumour location, its resectability and histology. As a group, however, the survival rate of childhood brain tumors has improved in recent years, resulting in an increased number of survivors returning to school and reintegrating into their communities. Survival for many of them, however, has also come with severe costs such as neurocognitive and academic difficulties. Cognitive rehabilitation strategies to address these deficits have been a major focus of recent research. Evidence is now also mounting for social competence deficits among this population which may persist into late adolescence and adulthood, thereby negatively affecting long-term survivorship. Thus, there is an urgency to identify psychosocial interventions, such as social skills programs, that can reduce the social competence deficits in childhood brain tumor survivors and, therefore, modify the course of these outcomes to ensure that survivors thrive and become productive members of society. To date, no rigorous social skills intervention trials have been undertaken to address the social difficulties of these survivors. The current proposal is the first study that aims to address this gap by evaluating the efficacy of an innovative, manualized, social skills intervention program developed for this population using a multi-centre Randomized Control Trial (RCT).

DETAILED DESCRIPTION:
Children and adolescents who are treated for brain tumours are faced with a variety of problems that affect the way they live their lives: one of the biggest problems is limited contact with friends and peers. This study aims to help kids and teens deal with this problem. The purpose of this study is to give kids who are treated for brain tumors opportunities to meet with other kids with similar experiences by participating in one of two social skills groups to improve how they related to one another. Investigators are assessing if these programs are beneficial to kids who have had brain tumours and which group is best. Kids will be assigned randomly to one of two groups. In both groups kids will meet with the other participants and with the facilitators for two hours once a week for 8 weeks. Kids in both groups will have introductions, group rules and group purpose (learn to relate with one another) through fun with games and arts and crafts. In one group, the games and crafts will be used for learning social skills. In the other group, arts and crafts and playing will be the focus of the activities, with the goal for each session determined by creating a craft or playing a game where everyone can win. One parent and all kids will complete questionnaires before the group starts, after the last group session as well as 6 months following the group. The questionnaires will ask questions about feeling, actions and getting along with others. Investigators also plan to visit the child's school so that the child, classmates and teachers will fill out questionnaires about friendships.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a brain/spinal tumour
2. off treatment for at least 3 months or on maintenance chemotherapy but medically stable, e.g., low grade gliomas
3. between 8 and 16 years of age at the time of enrollment
4. have sufficient fluency in English for active group participation
5. attending school regularly and in a regular classroom for at least 50% of a school day

Exclusion Criteria:

1. Severe cognitive deficits, as defined by enrollment in full-time special classroom, which will prevent them from participating fully
2. a diagnosis of conduct disorder or any other condition that may interfere with group activities. Survivors and parents who have some difficulties reading (i.e., English is their second language) will be assisted by a research assistant (RA) in completing the questionnaires.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2012-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Parent-rated social skills - assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  Measured by Social Skills Rating System (SSRS)[37]. The SSRS is a standardized instrument that has parent, teacher and child versions.
Child-rated social skills -- assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  Measured by Social Skills Rating System (SSRS)[37]. The SSRS is a standardized instrument that has parent, teacher and child versions.

SECONDARY OUTCOMES:
Quality of life ratings - general, parental assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  Quality of Life Inventory - PedsQL, generic[38] - Parent report
Quality of life ratings - general, child assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  Quality of Life Inventory - PedsQL, generic[38] - Child self-report
Quality of life ratings - brain tumour module, parent assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  Quality of Life Inventory - PedsQL, Brain Tumour Module[38] - parent report
Quality of life ratings - brain tumour module, child assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  Quality of Life Inventory - PedsQL, Brain Tumour Module[38] - Child self-report
Child's social functioning - assessment of change across three time points | day 1, 8 weeks later, and 6 months after day 1
  subscale of the Behavior Assessment System for Children-Second Edition, BASC-2, completed by parents

CONTACTS AND LOCATIONS:
Overall Officials: Maru Barrera, MD, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - Alberta Childrens Hospital, Calgary, Alberta
  - BC Women and Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Background] Butler RW, Mulhern RK. Neurocognitive interventions for children and adolescents surviving cancer. J Pediatr Psychol. 2005 Jan-Feb;30(1):65-78. doi: 10.1093/jpepsy/jsi017. PMID 15610986
- [Background] Reddick WE, White HA, Glass JO, Wheeler GC, Thompson SJ, Gajjar A, Leigh L, Mulhern RK. Developmental model relating white matter volume to neurocognitive deficits in pediatric brain tumor survivors. Cancer. 2003 May 15;97(10):2512-9. doi: 10.1002/cncr.11355. PMID 12733151
- [Background] Copeland DR, deMoor C, Moore BD 3rd, Ater JL. Neurocognitive development of children after a cerebellar tumor in infancy: A longitudinal study. J Clin Oncol. 1999 Nov;17(11):3476-86. doi: 10.1200/JCO.1999.17.11.3476. PMID 10550145
- [Background] Butler RW, Copeland DR. Attentional processes and their remediation in children treated for cancer: a literature review and the development of a therapeutic approach. J Int Neuropsychol Soc. 2002 Jan;8(1):115-24. PMID 11843068
- [Background] Radcliffe J, Bennett D, Kazak AE, Foley B, Phillips PC. Adjustment in childhood brain tumor survival: child, mother, and teacher report. J Pediatr Psychol. 1996 Aug;21(4):529-39. doi: 10.1093/jpepsy/21.4.529. PMID 8863462
- [Background] Vannatta K, Gartstein MA, Short A, Noll RB. A controlled study of peer relationships of children surviving brain tumors: teacher, peer, and self ratings. J Pediatr Psychol. 1998 Oct;23(5):279-87. doi: 10.1093/jpepsy/23.5.279. PMID 9782676
- [Background] Schulte F, Barrera M. Social competence in childhood brain tumor survivors: a comprehensive review. Support Care Cancer. 2010 Dec;18(12):1499-513. doi: 10.1007/s00520-010-0963-1. Epub 2010 Aug 1. PMID 20680353
- [Background] Barrera M, Shaw AK, Speechley KN, Maunsell E, Pogany L. Educational and social late effects of childhood cancer and related clinical, personal, and familial characteristics. Cancer. 2005 Oct 15;104(8):1751-60. doi: 10.1002/cncr.21390. PMID 16130127
- [Background] Zebrack BJ, Gurney JG, Oeffinger K, Whitton J, Packer RJ, Mertens A, Turk N, Castleberry R, Dreyer Z, Robison LL, Zeltzer LK. Psychological outcomes in long-term survivors of childhood brain cancer: a report from the childhood cancer survivor study. J Clin Oncol. 2004 Mar 15;22(6):999-1006. doi: 10.1200/JCO.2004.06.148. PMID 15020603